CLINICAL TRIAL: NCT07044947
Title: Non-interventional Real-World Study of Oteseconazole in the Treatment of Vulvovaginal Candidiasis
Brief Title: Oteseconazole in the Treatment of Adults With Vulvovaginal Candidiasis（VVC）
Acronym: VVC
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Qinping Liao, Chief physician, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: MA-VVC-RWS-002
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — VT-1161

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Oteseconazole: Subjects with SVVC will be treated with 600 mg (150 mg per capsule) on D1, 450 mg on D2
  Interventions: Drug: Oteseconazole (VT-1161) 150mg capsule

INTERVENTIONS:
Drug: Oteseconazole (VT-1161) 150mg capsule — Subjects with SVVC will be treated by Oteseconazole with 600 mg (150 mg per capsule) on D1, 450 mg on D2

SUMMARY:
Oteseconazole is a novel, oral, highly selective inhibitor of fungal CYP51. Oteseconazole showed statistically significant and clinically meaningful treatment of severe VVC and was generally tolerated. The trial is a national multi-center, non-interventional observational real-world study, aiming to evaluate the effecacy and safety of oteseconazole in the treatment of patients with VVC. This study will include patients with severe vulvovaginal candidiasis (SVVC) . It is divided into prospective and retrospective parts.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, female; vulvovaginal signs and symptoms (VSS) score ≥7; Plan to use oteseconazole monotherapy or combination therapy

Exclusion Criteria:

* Evidence has shown that the patient whohas been pregnant or lactating; Patients who are participating in or planning to participate in other interventional clinical studies; Other situations determined by the researcher as unsuitable for inclusion in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 3000
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2027-08-10 (Estimated); Study Completion 2030-08-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects achieving clinical cure at 6-month, | 6-month after the end of treatment
  clinical cure，defined as the absence of signs and symptoms of VVC

SECONDARY OUTCOMES:
The proportion of patients with clinical recurrence within 1-month, 12-month, 24-month and 36-month after treatment with Oteseconazole | 1-month, 12-month, 24-month and 36-month after the end of treatment
The time of the first clinical recurrence of VVC during the follow-up period | From enrollment to the end of treatment for 3 years"
Adverse events and serious adverse events from the time of signed consent to the end of the study | From enrollment to the end of treatment at 3 years